CLINICAL TRIAL: NCT03308240
Title: Magic Therapy to Relieve Pediatric Patient Anxiety and Improve the Hospitalization Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Maribeth Chitkara, Associate Professor of Clinical Pediatrics, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1037793-2
Record Dates: First submitted 2017-09-28; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Anxiety
Keywords: Magic; Anxiety; Pediatric
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two groups will be studied: an experimental group (patient and caregiver) receiving one magic therapy session within the hospitalization period and a control group (patient and caregiver) who will receive standard child life therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magic Therapy Group (Experimental): Medical student magicians who have completed MagicAid training will provide the therapy.
  Three or four tricks will be performed per patient at the discretion of the magician to cater to patient age and cognition capabilities. Patients in the experimental group may be given the opportunity to learn a magic trick that has been presented to them as well.
  Interventions: Behavioral: Magic Therapy
- Standard Child Life Therapy Group (No Intervention): Stony Brook Child Life Specialists will provide standard therapies available to all patients, such as pet therapy, art therapy, music therapy.

INTERVENTIONS:
Behavioral: Magic Therapy — As described in the arm description
  Arms: Magic Therapy Group

SUMMARY:
This study will assess the efficacy of magic therapy services in relieving pediatric patient anxiety and parent anxiety in an inpatient setting. It will also measure family satisfaction with child life services during the hospital visit and health professional opinions regarding such a therapy in an inpatient setting. The primary evaluation method will be through surveys. No prior investigations have studied using magic therapy as a primary tool to improve the psychological well-being of pediatric patients over the span of an inpatient hospitalization. Study and improvement of magic therapy services provides an evidence-based approach to improve pediatric patient psychological well-being, assist physicians in obtaining pediatric patient cooperation with procedures, and improving the hospitalization experience for the family of hospitalized pediatric patients.

DETAILED DESCRIPTION:
The use of magic in healthcare has been described across a variety of settings. Several peer-reviewed publications have described the use of magic to help encourage the recovery of motor skills 2. Green et al. reported that after the completion of an intense 2-week magic-theme summer camp, patients with spastic hemiplegia significantly increased the usage of their affected hand 3. Another investigation sought to study if magic could be used to aid in communication with mentally-disabled children 4. This study concluded that magic was effective in building trust, improving the subjects' self-esteem, and enriching their interpersonal skills.

Magic has also been partially studied in a surgical context for relieving perioperative anxiety. One study sought to evaluate the efficacy of clowns (whose performance included magic tricks) in relieving perioperative anxiety 5. Patients that were undergoing surgical procedures were placed in either a clown group or non-clown group. These patients were not grouped based on surgical procedures, and patients were included that were undergoing one of ten different surgeries. Anxiety levels of the pediatric patients were measured in the waiting room and induction room immediately prior to anesthesia administration. Additionally, parent state and trait anxiety was measured during their child's induction using the State-Trait Anxiety Inventory (STAI). Health professionals involved in the surgeries were also questioned using a questionnaire developed by the authors to obtain health providers' opinion regarding the presence of clowns as administered in the study. Moreover, clowns filled out a self-evaluation form regarding how they believed their interaction with the child went prior to the surgery. The authors found that the clown group displayed decreased anxiety during anesthesia induction but not in the waiting room. They also documented that health professionals believed the clowns benefitted the child, but at the same time, a majority of the staff discouraged continuance of the program due to interference with operating room procedures.

This study will assess the efficacy of magic therapy services in relieving pediatric patient anxiety and parent anxiety in an inpatient setting. It will also measure family satisfaction with child life services during the hospital visit and health professional opinions regarding such a therapy in an inpatient setting. The primary evaluation method will be through surveys. No prior investigations have studied using magic therapy as a primary tool to improve the psychological well-being of pediatric patients over the span of an inpatient hospitalization. Study and improvement of magic therapy services provides an evidence-based approach to improve pediatric patient psychological well-being, assist physicians in obtaining pediatric patient cooperation with procedures, and improving the hospitalization experience for the family of hospitalized pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* All 5-18 year-old patients that are admitted to the general pediatric inpatient pediatric unit at Stony Brook Children's
* All Caregivers of patients admitted to the general pediatric inpatient pediatric unit at Stony Brook Children's
* All medical professionals present on the pediatric inpatient unit at Stony Brook Children's during magic and child life service therapy.

Exclusion Criteria:

* Patients/caregivers who are not able to speak/read English
* Patients under the age of 5 years, as the instruments to be used to measure anxiety have not been validated in this age group.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-07-26 (Estimated); Study Completion 2018-07-26 (Estimated)

PRIMARY OUTCOMES:
To assess the therapeutic benefits of magic therapeutic intervention and impact on patient anxiety age 5-13 years. | 1-2 days per patient during course of hospitalization
  The Venham Picture Test (VPT) will be administed pre- and post-therapies (magic and standard child life therapies) to patients aged 5-13 to measure anxiety levels. The VPT is a measure of childhood state anxiety that has been validated for use in children aged 3-13 (Venham, Bengston, & Cipes, 1979). It has a series of pictures of faces expressing escalating levels of paint/anxiety.
To assess the therapeutic benefits of magic therapeutic intervention and impact on pediatric patient anxiety age 5-16 years. | 1-2 days per patient during course of hospitalization
  The Facial Image Scale will be administered pre- and post-therapies (magic and standard child life services) to children abed 5-16. The Facial Image Scale is a validated too that utilizes a series of five faces depicting faces ranging in expression from very happy to very unhappy (Buchanan & Niven, 2002). Children are asked at a specific time, which face they feel like at the moment. This scale has been used and validated in children aged 3-18.
To assess the therapeutic benefits of magic therapeutic intervention and impact on patient (age 5-16) and caregiver anxiety. | 1-2 days per patient during course of hospitalization
  The 6-item State-Trait Anxiety Inventory (STAI) is a validated tool which will be used to measure anxiety pre- and post-therapies (magic and standard child life therapies) for pediatric patients 5-16 years of age, and for caregivers of patients (Marteau & Bekker, 1992; Thanh Nhan Nguyen, Nilsson, Hellström, & Bengtson, 2010). This scale has also been validated in children from age 5-16 (Apell, Paradi, Kokinsky, Nilsson, & Kokinsky, 2011).

SECONDARY OUTCOMES:
To determine medical professional opinions regarding magic therapeutic services as offered at Stony Brook Children's Hospital. | One year, duration of patient/caregiver couplet enrollment
  Medical professionals will receive a questionnaire adapted from a prior study to assess their opinions regarding magic as a therapeutic intervention in an inpatient setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No